CLINICAL TRIAL: NCT07058818
Title: Tailored Resistance Training After Adverse Pregnancy Outcomes
Acronym: RT after APOs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Women's Health Innovation Fund (Unknown)
Responsible Party: Principal Investigator, Abbi Lane, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HUM00266890
Record Dates: First submitted 2025-06-11; First posted 2025-07-10 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Postpartum; Adverse Pregnancy Outcomes
Keywords: resistance training; postpartum health; adverse pregnancy outcomes
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Resistance training
  Interventions: Behavioral: Resistance training

INTERVENTIONS:
Behavioral: Resistance training — Full-body physical therapy and resistance training intervention

SUMMARY:
Approximately 7-10 postpartum people with recent adverse pregnancy outcomes (APOs: preeclampsia, gestational diabetes, hypertensive disorders of pregnancy, fetal growth restriction or low birth weight baby, or preterm birth) will be invited to complete 4 weeks of a resistance training intervention, including associated incentives, communication, and marketing materials.

DETAILED DESCRIPTION:
People who had APOs have a higher risk of heart disease and diabetes in the future. Resistance training might help lower risk of heart disease and diabetes in people who had APOs, but it can be difficult for postpartum people to perform exercise as they are juggling demands of a new baby and healing from pregnancy and child birth. The goal of this project is to find an exercise plan that works for individuals who recently gave birth. This study will determine whether a resistance training intervention co-designed by researchers and postpartum individuals is do-able for individuals who recently had APOs.

Participants in this trial will have height and weight measured. One exercise session, including a warm-up, resistance training, and cool-down with stretching will be completed in the School of Kinesiology at the University of Michigan. Then participants will receive an exercise program to perform over the next 4 weeks. An exercise session at around the midpoint of the program will be supervised by a trainer as a check point. They will receive a text or email message every day for those 4 weeks asking them to reply and tell the study team if they did the resistance training and if they did the program as it was written (as prescribed).

A few survey questions about participants mood regarding physical activity before and after exercise and belief in the ability to continue to exercise at the beginning and end of the intervention will be asked. Some questions regarding what participants thought about the marketing materials and the exercise program in general will be asked at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Had a single baby in your most recent pregnancy
* Are 18-45 years old
* Are 3-15 months postpartum
* Are not currently pregnant
* Had an adverse pregnancy outcome/medical complication in your most recent pregnancy, including preeclampsia, gestational diabetes, hypertensive disorders of pregnancy, fetal growth restriction or low birth weight baby, or preterm birth
* Your doctor told you that you are able to participate in exercise
* Are not currently meeting national physical activity guidelines, defined as 150 min/wk of aerobic exercise and 2 resistance training sessions/wk
* Can attend a visit at the University of Michigan's School of Kinesiology Building
* Are willing to perform resistance exercise twice a week for 4 weeks
* Are willing to receive and respond to a daily message sharing whether you completed resistance exercise that day and completed it as recommended

Exclusion criteria:

* Had a multiple birth (twins, triplets, etc) in your most recent pregnancy
* Are <18 or >45 years old
* Are <3 months or >15 months past your last birth
* Are currently pregnant
* Are unable to exercise or have been told by a healthcare provider not to exercise
* Are currently meeting national physical activity guidelines, defined as 150 min/wk of aerobic exercise and 2 resistance training sessions/wk
* Did not have an adverse pregnancy outcome, including preeclampsia, gestational diabetes, hypertensive disorders of pregnancy, fetal growth restriction or low birth weight baby, or preterm birth, in your most recent pregnancy
* Are unable to attend a study visit at the University of Michigan's School of Kinesiology Building
* Are not willing to perform 4 weeks of resistance training
* Are not willing to receive and send daily messages

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Adherence | 4 weeks
  Proportion of prescribed resistance exercise sessions completed
Compliance | 4 weeks
  Proportion of prescribed resistance exercise sessions completed as prescribed/directed

SECONDARY OUTCOMES:
Self-efficacy (assessed with validated survey) | 4 weeks
  Exercise self-efficacy survey
Physical activity enjoyment (assessed with validated survey) | 4 weeks
  Enjoyment questionnaire

OTHER OUTCOMES:
Opinions of exercise program | 4 weeks
  Program feedback provided during a semi-structured interview at the end of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Abbi Lane, PhD, Principal Investigator — University of Michigan
Locations (1):
- School of Kinesiology, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
The dataset will be small, and minimal data will be collected. It will be stored only at Michigan.